CLINICAL TRIAL: NCT06537765
Title: Combined Effect of Therapeutic Ultrasound and Trans Cutaneous Electrical Nerve Stimulation on Endometriosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Mohammed Ibrahim Mohammed Derwa, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012/003874
Record Dates: First submitted 2024-07-30; First posted 2024-08-05 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Ultrasonic Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapeutic ultrasound (US) Group (Experimental): It will include 15 women, who will receive their hormonal treatment as prescribed by the gynecologist in addition to, Therapeutic US, 3 sessions, per week for eight weeks.
  Interventions: Drug: Medical treatment; Device: Therapeutic ultrasound (US)
- Transcutaneous Electrical Nerve Stimulation (TENS) Group (Experimental): It will include 15 women, who will receive their hormonal treatment as prescribed by the gynecologist in addition to, TENS therapy, 3 sessions, per week for eight weeks.
  Interventions: Drug: Medical treatment; Device: Transcutaneous electrical nerve stimulation (TENS)
- US + TENS Group (Experimental): It will include 15 women, who will receive their hormonal treatment as prescribed by the gynecologist in addition to, both Therapeutic US and TENS therapy, 3 sessions, per week for eight weeks.
  Interventions: Drug: Medical treatment; Device: Therapeutic ultrasound (US); Device: Transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Drug: Medical treatment — All women with endometriosis in all groups (A, B, & C) will receive their medical treatment as prescribed by the gynecologist.
Device: Therapeutic ultrasound (US) — Women will be asked to assume supine lying position, and the lower abdomen will be cleaned thoroughly with alcohol and dried well thereafter. Ultrasound gel will be distributed over the lower abdomen .The device will be adjusted to Frequency of 1MHz, Mode: continuous wave, Intensity: 1.5W/cm, duration of treatment: 15 minutes for the treatment site, then the skin will be cleaned again to remove ultrasound gel.
  Arms: Therapeutic ultrasound (US) Group; US + TENS Group
Device: Transcutaneous electrical nerve stimulation (TENS) — TENS electrodes will be placed on specific acupuncture points for women in supine position. These points include VB29, ST36, CV6, CV4, LV3, KD3, SP6, and SP9. The treatment aims to improve blood circulation, remove adhesions, regulate menstrual activity and hormones, and prevent new adhesions and menstrual reflux in endometriosis patients.
  Arms: Transcutaneous Electrical Nerve Stimulation (TENS) Group; US + TENS Group

SUMMARY:
This study will be conducted to investigate the combined effect of therapeutic ultrasound and transcutaneous electrical nerve stimulation (TENS) on relieving adhesions and pain related to endometriosis.

DETAILED DESCRIPTION:
Endometriosis affects 10-15% of reproductive-age women, causing pelvic pain and infertility. While laparoscopy is the primary treatment, it has risks. Medications are also used but often have side effects. Complementary therapies like acupuncture, yoga, and physical therapy modalities show promise. Therapeutic ultrasound has demonstrated effectiveness in managing chronic pain and adhesions associated with endometriosis. Transcutaneous electrical nerve stimulation (TENS) has shown positive results in pain relief and potentially improving uterine conditions for implantation. This study aims to investigate the combined effect of therapeutic ultrasound and TENS on endometriosis-related adhesion and pain, providing valuable information for physical therapists in treating this condition.

ELIGIBILITY:
Inclusion Criteria:

* Forty-five women clinically diagnosed by the gynecologist with endometriosis will be included in the study.
* Abdominal wall endometriosis will be diagnosed via Color Doppler ultrasonography.
* Their ages will range from 25 to 35 years old.
* Their body mass index (BMI) will be ranged from 25 to 35 Kg/m2.
* All patients have reported mild to moderate endometriosis symptoms such as (chronic pelvic pain (CPP), dysmenorrhea, dyspareunia, pain with bowel movements and urination and excessive bleeding) as recorded by Endometriosis Health profile questionnaire (EHP30).
* All patients use continuous hormonal treatment for at least 3 months.

Exclusion Criteria:

* Severe endometriosis which is diagnosed by the gynecologist.
* Pregnancy, peacemaker, epilepsy, cardiac arrhythmia, cancer, acute inflammatory pelvic disease.
* Use of injectable hormonal therapy within the previous 6 weeks.
* Patients with contraindication of ultrasound (Patients with reduced sensation to pain and/or heat, local malignancy, local acute infection and over areas of thrombosis or other vascular abnormalities).
* Cognitive deficiency and difficulty to understand instructions or use the instruments.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of adhesion size | 8 weeks
  New Color Doppler Ultrasound scanner will be used in the study to assess adhesion size for all women with endometriosis in all groups (A, B, & C) before and after the study, and this procedure will be applied by the gynecologist.
The McGill pain questionnaire (MPQ) | 8 weeks
  The pain intensity for all groups (A, B, & C) will be assessed using the McGill Pain Questionnaire (MPQ) before and after the treatment program. The MPQ is a comprehensive tool that evaluates various dimensions of a patient's pain experience through three parts. The first part includes an anatomical drawing where the patient marks the location of their pain. The second part is a Verbal Descriptor Scale (VDS) for the patient to indicate the intensity of their current pain. The third part is an inventory of 72 descriptive adjectives to detail the pain further. The MPQ measures three key aspects: (1) the pain rating index, which assigns numerical values to each word descriptor, (2) the number of words chosen, and (3) the present pain intensity on a 1-5 scale (1 for mild, 2 for discomforting, 3 for distressing, 4 for horrible, and 5 for excruciating).
The Endometriosis Health profile (EHP30) questionnaire | 8 weeks
  The Endometriosis Health profile (EHP30) questionnaire will be used to assess symptoms of endometriosis in all groups (A, B & C) before and after the end of treatment program. It is self-reporting instrument that contains a core questionnaire consisting of 30 items assessing five dimensions. The five dimensions included pain, control and impotence, emotional well-being, social support, and self
  -image. Each scale is converted into a score from 0 to 100, with a lower score representing a better quality of life.

SECONDARY OUTCOMES:
The Health-related quality of life (HRQOL-36) questionnaire | 8 weeks
  The Health-related quality of life (HRQOL-36) questionnaire will be used to assess health related quality of life for all women with endometriosis in all groups (A, B & C) before and after the end of treatment program. It is a reliable and validated disease specific questionnaire with 36 questions that encompass five core scales: pain, control and powerlessness, emotional well-being, social support, and self- image. Questions are asked regarding endometriosis and are answered on a 5-points Likert scale, where 0=never, 1=rarely, 2=sometimes, 3=often, and 4=always. Raw scores for the questions within a scale are summed and transformed to a 0-100 scale, with higher scores indicating worse health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Soheir El-Kosery, PhD, Study Chair — Professor of Physical Therapy for Women's Health